CLINICAL TRIAL: NCT05594186
Title: Nonsurgical Management of Cesarean Scar Niche Related Abnormal Uterine Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saudi German Hospital - Madinah (Other)
Responsible Party: Principal Investigator, Islam Mohamed Magdi Ammar, Consultant and associate Professor of Obstetrics and Gynecology, Saudi German Hospital - Madinah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGHM-FEB2019-OBGYN
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Intermenstrual Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tranexamic acid (Active Comparator): Patients in group A, received Tranexamic acid 1300 mg (2 tablets of 650 mg) three times daily for 5 days starting from the first day of menses for 12 months.
  Interventions: Drug: Tranexamic acid, Oral contraceptive pills and the Levonorgestrel-releasing intrauterine system.
- Combined oral contraceptive pill (Active Comparator): Patients in group B, received combined oral contraceptive pill (OCP) once daily for 21 days (Desogestrel 150 micrograms/ Ethinylestradiol 30 micrograms, tablets), starting from the first day of menses, then to have a one-week pill free period to allow for a withdrawal bleed, and that was repeated for 12 cycles.
  Interventions: Drug: Tranexamic acid, Oral contraceptive pills and the Levonorgestrel-releasing intrauterine system.
- Tranexamic acid plus Combined oral contraceptive pill (Active Comparator): Patients in group C, received a combination of Tranexamic acid 1300 mg three times daily for 5 days, and a combined oral contraceptive pill once daily for 21 days (Desogestrel 150 micrograms/ Ethinylestradiol 30 micrograms, tablets), both starting from the first day of menses for 12 consecutive cycles.
  Interventions: Drug: Tranexamic acid, Oral contraceptive pills and the Levonorgestrel-releasing intrauterine system.
- Levonorgestrel-releasing intrauterine system (Active Comparator): Patients in group D, had the levonorgestrel-releasing intrauterine system inserted into the uterine cavity. The insertion was done by a skilled gynecologist as an outpatient procedure without anesthesia.
  Interventions: Drug: Tranexamic acid, Oral contraceptive pills and the Levonorgestrel-releasing intrauterine system.

INTERVENTIONS:
Drug: Tranexamic acid, Oral contraceptive pills and the Levonorgestrel-releasing intrauterine system. — Comparing three different nonsurgical management options for abnormal uterine bleeding caused by cesarean scar niche.

SUMMARY:
A study of the effect of three different nonsurgical methods for management of abnormal uterine bleeding caused by cesarean scar niche. The study was conducted at the Obstetrics and Gynaecology department of the Saudi German Hospital in Madinah- Saudi Arabia, during the period between March 2019 to October 2022. The study protocol was in accordance with the Helsinki declaration 1964 and the later amendments. A prospective approval was granted by the human research ethics committee of the hospital and the study participants have signed an informed consent.

DETAILED DESCRIPTION:
The study included 158 patients aged between 20 and 40 years who had a history of at least one caesarean delivery and presented with abnormal uterine bleeding in the form of postmenstrual spotting defined as bloody or brownish discharge of more than two days after the end of menstruation, with the total duration of (menses and spotting) of more than 7 days, or intermenstrual bleeding that starts after the end of the menses, who were diagnosed to have a caesarean scar niche by saline infusion sonography. Cesarean scar niche was defined as an anechoic triangular indentation at the site of the previous cesarean scar with a depth of at least 2 mm. Exclusion criteria were: pregnancy, desire for fertility within one year of enrolment in the study, any medical condition contraindicating the use of combined oral contraceptive pills, history of abnormal uterine bleeding dating before the last caesarean section, use of any hormonal treatment 3 months prior to enrolment, coagulopathy, and organic causes of bleeding like uterine fibroids, adenomyosis or endometrial hyperplasia. Saline infusion sonography was done, in which instillation of saline solution into the uterine cavity, enhanced the transvaginal ultrasonographic image by providing a sonolucent contrast medium to allow for better visualization and delineation of the defect. Evaluation was performed according to the 2019 modified Delphi procedure where the basic evaluation of CS niche included measurements of the length, depth and width of the defect, the residual myometrial thickness (RMT) and the adjacent myometrial thickness (AMT). All measurements were made in the sagittal plane except the width which was measured in the transverse plane. The 4.5 MHz endovaginal transducer (Canon Xario 200G Ultrasound, Japan) was used.

Using an Open Epi version 3.21 computer-based software, patients were divided into four groups (A, B, C and D). Patients in group A, received Tranexamic acid 1300 mg (2 tablets of 650 mg) three times daily for 5 days starting from the first day of menses for 12 months. Patients in group B, received combined oral contraceptive pill (OCP) once daily for 21 days starting from the first day of menses, then to have a one-week pill free period to allow for a withdrawal bleed, and that was repeated for 12 cycles. Patients in group C, received a combination of Tranexamic acid 1300 mg three times daily for 5 days, and a combined oral contraceptive pill once daily for 21 days, both starting from the first day of menses for 12 consecutive cycles. Patients in group D, had the levonorgestrel-releasing intrauterine system inserted into the uterine cavity. The insertion was done by a skilled gynecologist as an outpatient procedure without anesthesia. The possible long- and short-term side effects of the different interventions were carefully discussed with all patients, and those who were willing to participate had signed the informed consent before participation. The primary outcome was the improvement of postmenstrual spotting as reported by the patients in their menstrual diary at each of the follow up visits (three, six, nine and twelve months) after enrolment in the study.

The participants were asked to complete the menstrual diary card that was designed based on that used in the study of Johannes and colleagues in 1996. The illustrated symbols at the top of the card indicated the heaviness of menstrual bleeding (flooding, heavy, normal, light or spotting) and the names of the months were written on the left side of the card.

ELIGIBILITY:
Inclusion Criteria:

* The study included 158 patients aged between 20 and 40 years who had a history of at least one caesarean delivery and presented with abnormal uterine bleeding in the form of postmenstrual spotting defined as bloody or brownish discharge of more than two days after the end of menstruation, with the total duration of (menses and spotting) of more than 7 days, or intermenstrual bleeding that starts after the end of the menses, who were diagnosed to have a caesarean scar niche by saline infusion sonography. Cesarean scar niche was defined as an anechoic triangular indentation at the site of the previous cesarean scar with a depth of at least 2 mm. Saline infusion sonography was done, in which instillation of saline solution into the uterine cavity, enhanced the transvaginal ultrasonographic image by providing a sonolucent contrast medium to allow for better visualization and delineation of the defect. Evaluation was performed according to the 2019 modified Delphi procedure where the basic evaluation of CS niche included measurements of the length, depth and width of the defect, the residual myometrial thickness (RMT) and the adjacent myometrial thickness (AMT). All measurements were made in the sagittal plane except the width which was measured in the transverse plane. The 4.5 MHz endovaginal transducer was used.

Exclusion Criteria:

* Exclusion criteria were: pregnancy, desire for fertility within one year of enrolment in the study, any medical condition contraindicating the use of combined oral contraceptive pills, history of abnormal uterine bleeding dating before the last caesarean section, use of any hormonal treatment 3 months prior to enrolment, coagulopathy, and organic causes of bleeding like uterine fibroids, adenomyosis or endometrial hyperplasia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Improvement of post-menstrual spotting | 12 months
  Improvement of post-menstrual spotting as reported by the patients in their menstrual diary at each of the follow up visits (three, six, nine and twelve months) after enrolment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mohamed Magdi Ammar, M.D., Principal Investigator — Saudi German Hospital - Madinah
Locations (1):
- Saudi German Hospital, Al Madīnah, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No